CLINICAL TRIAL: NCT01500551
Title: A LONG-TERM, OPEN-LABEL FOLLOW-UP STUDY OF TOFACITINIB FOR TREATMENT OF JUVENILE IDIOPATHIC ARTHRITIS (JIA)
Brief Title: Long-Term Safety Study Of Tofacitinib In Patients With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3921145; JIA (Other: Alias Study Number); 2023-509651-14-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Arthritis; Pediatric; Long-term; JIA; CP-690,550; tofacitinib; Xeljanz
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tofacitinib (Experimental): All patients will be in tofacitinib treatment group.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib will be administered orally BID (twice daily) approximately 12 hours (±2 hours) apart, once in the morning and once in the evening, based on body weight for all subjects for all three index studies (A3921103, A3921104, and A3921165)
  5 mg BID Dose Level:
  Body Weight (Dose in tablet [mg BID] or solution [ml BID]) 5 - < 7 kg (2 mg or 2 ml) 7 - < 10 kg (2.5 mg or 2.5 ml) 10 - <15 kg (3 mg or 3 ml) 15 - <25 kg (3.5 mg or 3.5 ml) 25 - <40 kg (4 mg or 4 ml) >=40 kg (5 mg or 5 ml)
  Oral solution (1 mg/mL concentration) will be used for subjects weighing <40 kg. Oral tablets (5 mg) will be used for subjects weighing >=40 kg; subjects who are unable to swallow tablets will have the option of taking oral solution.
  Subjects will swallow study tablets whole and will not manipulate or chew tablets prior to swallowing.
  Other Names: CP 690,550, Xeljanz
Drug: Tofacitinib — For subjects rolling over from study A3921103 and actively participating in this study at the time of Protocol Amendment 6 and receiving a dosage of tofacitinib in accordance with the dosing scheme specified in Protocol Amendment 5, investigators will have the option of maintaining the subject's current dosage regimen from index study A3921103 (if the desired clinical response has been attained with no safety concern) or adjusting the dosage regimen in accordance with the dosing scheme specified in this section.
  Other Names: CP-690,550, Xeljanz

SUMMARY:
Evaluate long-term safety and tolerability of tofacitinib in patients with JIA, who have previously participated in tofacitinib JIA studies.

DETAILED DESCRIPTION:
This is a Phase 2/3, long term, open-label, follow-up study. Subjects will have previously participated in qualifying/index JIA studies of tofacitinib. Those who have already completed such participation and enroll outside the 14 day window following completion of the End of Study (EOS) Visit of the qualifying/index study will participate in a screening Visit to determine eligibility. A Baseline Visit will then occur within 28 days after the Screening Visit. For subjects who are completing participation in a qualifying study of tofacitinib and enrolling on the same day of the EOS Visit of the qualifying/index study, the EOS Visit of the qualifying/index study can be combined with the Screening and Baseline Visits for this study. The subjects who enroll within the 14 day window following completion of the EOS Visit of the qualifying/index study will participate in a combined Screening and Baseline Visit for this study. After the Baseline Visit, visits will occur at 1 month (1 month=30 days) and 3 months, then every 3 months thereafter as long as the subject remains in the study.

Approximately 340 participants are projected to enroll into this open label extension study after completing a qualifying/index study in the JIA program.

For subjects who entered this study from the A3921103 and A3921104 qualifying/index studies, their participation in this study ends after the first marketing approval of tofacitinib for the treatment of polyarticular course Juvenile Idiopathic Arthritis (pJIA) in any country. This study will end once the last subject, and all other subjects, who entered from index study A3921165 have completed approximately 1 year in this study, or after the first marketing approval of tofacitinib for the treatment of systemic JIA, whichever comes first.

The total duration of an individual subject's participation may vary depending upon when they enter the trial.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects with JIA aged from 2 to less than 18 years who met entry criteria for the qualifying/index study and in the opinion of the investigator have sufficient evidence of JIA disease activity to warrant use of tofacitinib as a DMARD. Subjects turning 18 years of age during participation in the qualifying/index study or subsequently will be eligible for participation in this study.
* The subject has discontinued disallowed concomitant medications for the required time prior to the first dose of study drug, as defined in Appendix 1, and is taking only those concomitant medications in doses and frequency allowed by the protocol.
* Fertile male subjects and female subjects of childbearing potential who are, in the opinion of the investigator, sexually active and at risk for pregnancy with their partner(s) must be using a highly effective method of contraception as outlined in this protocol throughout the study and for at least 28 days after the last dose of study medication.
* Subjects must have previously completed participation in a qualifying study of tofacitinib for the treatment of JIA. Subjects who have required earlier discontinuation of treatment in a qualifying study for reasons other than tofacitinib related serious adverse events may be eligible.

Exclusion Criteria:

* persistent oligoarthritis, and undifferentiated JIA.
* Infections:

  1. Chronic infections.
  2. Any infection requiring hospitalization, parenteral antimicrobial therapy or judged to be opportunistic by the investigator within the 3 months prior to the first dose of study drug.
  3. Any treated infections within 2 weeks of baseline visit.
  4. A subject known to be infected with human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus.
  5. History of infected joint prosthesis with prosthesis still in situ.
* History of recurrent (more than one episode) herpes zoster or disseminated (a single episode) herpes zoster or disseminated (a single episode) herpes simplex.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 302 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Standard laboratory safety data and adverse event (AE) reports. Body weight, height and Tanner Stages will collected to assess growth and physical development. | up to 8 years

SECONDARY OUTCOMES:
Physician global evaluation of disease activity at each visit. | up to 8 years
Number of joints with active arthritis at each visit. | up to 8 years
Number of joints with limitation of motion at each visit. | up to 8 years
Index of inflammation (C-reactive protein [CRP] and Erythrocyte Sedimentation Rate [ESR]) at each visit. | up to 8 years
Parent's Assessment of Physical Function (Childhood Health Assessment Questionnaire [CHAQ]Disability Index)at each visit. | up to 8 years
Parent's Assessment of Child's Arthritis Pain (Childhood Health Assessment Questionnaire [CHAQ] Discomfort Index, Visual Analog Scale [VAS])at each visit. | up to 8 years
Parent's Global Assessment of Overall Wellbeing (Childhood Health Assessment Questionnaire [CHAQ] subsection, Visual Analog Scale [VAS])at each visit. | up to 8 years
JIA American College of Rheumatology (ACR) response and occurrence of JIA ACR disease flare at each visit. | up to 8 years
JIA ACR Clinical Inactive Disease status and Clinical Remission on Medication at each visit. | up to 8 years
Change from baseline in Juvenile Arthritis Disease Activity Score (JADAS) 27- CRP and JADAS 27-ESR, and occurrence of JADAS minimum disease activity and inactive disease at each visit. | up to 8 years
In subjects with Enthesitis Related Arthritis (ERA): Change from baseline in the Tender Entheseal Assessment, Modified Schober's Test, Overall Back Pain and Nocturnal Back Pain responses at various visits. | up to 8 years
In subjects with psoriatic arthritis (PsA): Change from baseline in body surface area (BSA) affected by psoriasis and Physician's Global Assessment (PGA) of psoriasis) at various visits. | up to 8 years
In subjects with sJIA: "Absence of Fever", defined as absence of fever due to sJIA in the week preceding the assessment at each visit. | up to 8 years
Eligibility of tapering defined per protocol for corticosteroids | up to 8 years
Eligibility of tapering defined per protocol for methotrexate | up to 8 years
Eligibility of tapering defined per protocol for leflunomide | Up to 8 years
Eligibility of tapering defined per protocol for tofacitinib | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (104):
- United States (43):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Children'S Hospital, Loma Linda, California
  - Loma Linda University Clinical Trials Center, Loma Linda, California
  - Loma Linda University Eye Institute, Loma Linda, California
  - Loma Linda University General Pediatric Clinic - Meridian, Loma Linda, California
  - Pediatric Speciality Team Centers of LLU Children's Hospital (Rheumatology), Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Pediatric Speciality Team Centers of LLU Children's Hospital (Rheumatology), San Bernardino, California
  - Rady Children's Hospital Center for Pediatric Clinical Research, San Diego, California
  - Rady Children's Hospital Rheumatology Clinic, San Diego, California
  - Rady Children's Hospital San Diego- Education and Office Building, San Diego, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Rady Children's Research Pharmacy, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - IDS Pharmacy, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Center for Advanced Pediatrics, Atlanta, Georgia
  - AU Medical Center, Augusta, Georgia
  - Augusta University, Augusta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Tufts Medical Center - Floating Hospital for Children, Boston, Massachusetts
  - Explorer Clinic, University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cohen Children's Medical Center of New York, Lake Success, New York
  - Columbia University Medical Center-Herbert Irving Pavillion, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Pediatric Research, Charlotte, North Carolina
  - Levine Children's Specialty Center, Charlotte, North Carolina
  - Atrium Health- Investigational Drug Services, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Group, Dell Children's Medical Center, Austin, Texas
  - Texas Children's Hospital- Clinical Care Center, Houston, Texas
  - Texas Children's Hospital- Clinical Research Center, Houston, Texas
  - Texas Children's Hospital- Investigational Pharmacy, Houston, Texas
  - Texas Children's Hospital- Main Hospital, Houston, Texas
  - Texas Children's Hospital/Baylor College of Medicine- Feigin Center, Houston, Texas
  - Intermountain - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Argentina (3):
  - Instituto CAICI SRL, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Hospital Britanico de Buenos Aires, CABA
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - The Royal Children's Hospital, Parkville, Victoria
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven - Gasthuisberg, Leuven
- Brazil (7):
  - SER - Serviços Especializados em Reumatologia, Salvador, Estado de Bahia
  - CMIP - Centro Mineiro de Pesquisa Ltda, Juiz de Fora, Minas Gerais
  - Hospital Pequeno Príncipe Clinical Research Office, Curitiba, Paraná
  - Faculdade de Medicina da UNESP, Botucatu, São Paulo
  - Instituto de Puericultura e Pediatria Martagao Gesteira (IPPMG), Rio de Janeiro
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina, São Paulo
  - Instituto da Crianca do Hospital das Clinicas da FMUSP, São Paulo
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - McGill University Health Center, Glen Site, Montreal, Quebec
- China (3):
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - The Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Children's Hospital, Capital Medical University/Rheumatology Department, Beijing
- Germany (4):
  - PRI - Pediatric Rheumatology Research Institute GmbH, Bad Bramstedt
  - Hamburger Zentrum fur Kinder und Jugendrheumatologie, Hamburg
  - Asklepios Klinik Sankt Augustin GmbH, Sankt Augustin
  - St. Josef-Stift Sendenhorst, Sendenhorst
- India (4):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - Institute of Child Health, Kolkata, West Bengal
  - Institute of Post Graduate Medical Education and Research & SSKM Hospital, Kolkata, West Bengal
  - Sir Ganga Ram Hospital, New Delhi
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center - Pediatric Clinic, Kfar Saba
  - Chaim Sheba M.C Tel hashomer, Ramat Gan
- Mexico (5):
  - Clínica de Investigacion en Reumatologia y Obesidad, S.C., Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro de Alta Especialidad de Reumatología e Investigación del Potosí, S.C., San Luis de Potosí
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City
  - Unidad de Investigaciones Reumatologicas A.C., San Luis Potosí City
- Poland (4):
  - Wojewodzki Szpital Dzieciecy im. J. Brudzinskiego, Bydgoszcz
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im. Sw. Ludwika w Krakowie, Krakow
  - Klinika Kardiologii i Reumatologii Dzieciecej, Lodz
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
- Russia (8):
  - FSBEI HE BSMU MoH RF, Ufa, Bashkortostan Republic
  - Clinic of FSBEI HE BSMU MoH RF, Ufa, Bashkortostan Republic
  - Federal State Budgetary Scientific Institution, Moscow
  - FSAEI HE I.M. Sechenov First MSMU of Minzdrav of Russia (Sechenovskiy University), Moscow
  - FSAEI HE I.M. Sechenov First MSMU of Minzdrav of Russia (Sechenovskiy University),, Moscow
  - FSAI "NMRCCH" of MOH Russia, Moscow
  - FSBEI HE "St. Petersburg State Pediatric Medical University" of the Ministry of Healthcare, Saint Petersburg
  - State Budgetary Healthcare Institution of Samara Region "Tolyatti City Clinical Hospital #5", Tolyatti
- Narodny ustav reumatickych chorob, Piešťany, Slovakia
- South Africa (2):
  - Panorama Medical Centre, Panorama, CAPE TOWN
  - Durban International Clinical Research Site, Enhancing Care Foundation, Durban
- Spain (3):
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty, Ankara
  - Umraniye Training and Research Hospital, Istanbul
  - Istanbul Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi Cocuk Romatoloji Bolumu, Kadikoy / Istanbul
- Ukraine (3):
  - Communal Institution "Dnipropetrovsk Specialized Clinical Medical Center of Mother and Child n.a., Dnipro
  - Ivano-Frankivsk Regional Children's Clinical Hospital, Ivano-Frankivsk
  - Communal Non-profit Enterprise, Vinnytsia
- Birmingham Woman's and Children's NHS Foundation Trust, Birmingham, WEST Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brunner HI, Akikusa JD, Al-Abadi E, Bohnsack JF, Boteanu AL, Chedeville G, Cuttica R, De La Pena W, Jung L, Kasapcopur O, Kobusinska K, Schulert GS, Neiva C, Rivas-Chacon R, Rizo Rodriguez JC, Vazquez-Del Mercado M, Wagner-Weiner L, Weiss JE, Wouters C, Posner H, Wouters A, Chang C, White C, Kanik K, Liu S, Martini A, Lovell DJ, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO) and Pediatric Rheumatology Collaborative Study Group (PRCSG). Safety and efficacy of tofacitinib for the treatment of patients with juvenile idiopathic arthritis: preliminary results of an open-label, long-term extension study. Ann Rheum Dis. 2024 Oct 21;83(11):1561-1571. doi: 10.1136/ard-2023-225094. PMID 38849152
- [Derived] Chang C, Vong C, Wang X, Hazra A, Diehl A, Nicholas T, Mukherjee A. Tofacitinib pharmacokinetics in children and adolescents with juvenile idiopathic arthritis. CPT Pharmacometrics Syst Pharmacol. 2024 Apr;13(4):599-611. doi: 10.1002/psp4.13104. Epub 2024 Jan 31. PMID 38298058
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921145